CLINICAL TRIAL: NCT05752812
Title: The HELPP Score: A Pretreatment Prognostic Score to Predict Survival and Patterns of Recurrence in Localized Non-Metastatic Pancreatic Cancer - a Multicenter Prospective Validation Study
Brief Title: The HELPP Score: A Pretreatment Score to Predict Survival in Pancreatic Cancer
Status: Recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Oliver Strobel, MD MBA, Prof. Dr. , MBA, Medical University of Vienna
Other Study IDs: MUVienna HELPP
Record Dates: First submitted 2023-02-21; First posted 2023-03-03 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: Pancreatic Ductal Adenocarcinoma; Pancreatic Resection; Preoperative Prognostic Score; Localized Non-Metastatic Pancreatic Ductal Adenocarcinoma; Recurrence
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to validate a pretreatment prognostic score (Heidelberg Prognostic Pancreatic Cancer Score - HELPP) in patients with pancreatic ductal adenocarcinoma.

The main questions it aims to answer are:

* Is the HELPP score able to predict median overall survival in a prospective multi-institutional cohort of patients with pretherapeutic localized non-metastatic pancreatic cancer?
* Is the HELPP score able to predict median recurrence-free survival and patterns of recurrence after resection of pancreatic cancer?

DETAILED DESCRIPTION:
Accurate pretreatment staging and subsequent prediction of prognosis in pancreatic ductal adenocarcinoma (PDAC) is challenging due to subclinical micrometastasis as well as variations in tumor biology. Moreover, patients with non-metastasized localized PDAC are increasingly treated with neoadjuvant chemotherapy prior to resection.

The investigators recently developed a preoperative prognostic score to predict postoperative outcomes based on routine laboratory biomarkers and the American Society of Anesthesiologists (ASA) score, the HELPP score (Heidelberg Prognostic Pancreatic Cancer Score). Based on a large retrospective analysis of 1197 patients and an external validation cohort the HELPP score was able stratify patients based on expected survival only utilizing routinely available preoperative data. However, prospective validation is currently lacking.

This multi-site prospective observational study aims to prospectively validate the HELPP score in the clinical scenarios described above. Additionally, it aims to investigate its utility regarding median recurrence-free survival and patterns of recurrence. The study includes all consecutive patients with PDAC undergoing exploration (without or without neoadjuvant treatment) with the aim of resection within a timeframe of 12 months (all-comers concept, snapshot study).

The parameters on which the score is based on are routinely available to hospitals worldwide. Simplicity of the grading system facilitates implementation in daily clinical practice. This score could potentially help tailor treatments, aid in patient stratification in clinical trials, and provide new insights into tumor biology.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* fit to undergo elective pancreatic resection or palliative therapy
* localized non-metastatic pancreatic ductal adenocarcinoma
* informed consent provided

Exclusion Criteria:

* patients with a diagnosis other than pancreatic ductal adenocarcinoma on histopathology
* missing informed consent
* missing mandatory pretreatment laboratory values
* missing mandatory pretreatment clinicopathologic data
* patients receiving surgery for peripancreatic cancer
* incomplete follow-up records
* follow-up < 24 months
* pregnancy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients presenting with localized non-metastatic pancreatic ductal adenocarcinoma undergoing treatment (upfront resection, resection after neoadjuvant therapy, or palliative therapy) at participating centers.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Median overall survival | Date of diagnosis to date of death; assessed up to 60 months
  Median overall survival from the time of diagnosis with pancreatic ductal adenocarcinoma to time of death due to any cause.

SECONDARY OUTCOMES:
Recurrence-free survival | Date of surgery to date of the first evidence of recurrent disease; assessed up to 60 months
  Median recurrence-free survival from the date of potentially curative pancreatic surgery for pancreatic ductal adenocarcinoma until detection of the first evidence of recurrent disease either based on cross-sectional imaging or cytology/histology.
Patterns of recurrence | Date of surgery to date of the first evidence of recurrent disease; assessed up to 60 months
  Patterns of recurrence either based on cross-sectional imaging or cytology/histology after potentially curative pancreatic surgery of pancreatic ductal adenocarcinoma. The location of recurrence will be defined based on the first site of recurrence. Only the first site of recurrence will be considered.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Strobel, MD MBA, Study Director — Medical University Vienna
Locations (1):
- Department of General Surgery, Division of Visceral Surgery, Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hank T, Hinz U, Reiner T, Malleo G, Konig AK, Maggino L, Marchegiani G, Kaiser J, Paiella S, Binco A, Salvia R, Hackert T, Bassi C, Buchler MW, Strobel O. A Pretreatment Prognostic Score to Stratify Survival in Pancreatic Cancer. Ann Surg. 2022 Dec 1;276(6):e914-e922. doi: 10.1097/SLA.0000000000004845. Epub 2021 Mar 4. PMID 33914468